CLINICAL TRIAL: NCT01943266
Title: Use of Indicator Amino Acid Oxidation Technique to Determine Protein Requirement of Elderly Male Subjects 65-75 Yrs Old.
Brief Title: Determination of Protein Requirement in Elderly Male Subjects 65-75 Yrs Old.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr. Paul Pencharz, Senior Scientist, The Research Institute, Hospital for Sick Children, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0019850580-C
Record Dates: First submitted 2013-08-16; First posted 2013-09-16 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Healthy Males 65-75 Yrs Old

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- protein intake (Experimental): protein intake randomly fed from deficient to excess
  Interventions: Dietary Supplement: protein intake

INTERVENTIONS:
Dietary Supplement: protein intake — on the study day, the diet will be provided as free amino acids,with calories made up by a liquid diet and protein free cookies. Protein intake will be varied at 0.2, 0.5, 0.7, 0.9, 1.0, 1.2, 1.5, 1.8, and 2.0 g.kg/day

SUMMARY:
Minimal data are available on protein requirements throughout the lifespan. Currently available recommendations are based on nitrogen balance data. The limitations of the nitrogen balance method have been well described. Importantly, nitrogen balanced underestimates requirements.

The current dietary reference intakes (DRI) requirement for healthy adult males is based on the reanalysis of the nitrogen balance date from Young and Scrimshaw. This data was reanalyzed statistically by Rand et al. and he concluded that the protein requirement of healthy adults was 0.65 and 0.83 (mean and RDA) g/kg/day of good quality protein. Using indicator amino acid oxidation (IAAO), our group estimated the protein requirement of young men (mean age 27 years) to be 0.93 and 1.2 g/kg/day (mean and RDA).

Currently there are no studies on protein requirement in the elderly. In a recent nutrition survey conducted by national health and nutrition examination survey (NHANES), the authors concluded that adults between the ages of 51 - 70 years old consumed an average on 1.0 g/kg/day (ideal body weight) of protein which represents about 15 % of calories. Depending on the calculations used for ideal body weight some older adults could be getting higher or lower than requirement. There is no scientifically derived protein estimate for older adults. Therefore there is a need to measurer protein requirement in that population.

The goal of this study therefore is to measure the protein requirement of male elderly subjects between the ages of 65 - 75 years using the IAAO technique.

ELIGIBILITY:
* Inclusion Criteria:

  1. Healthy elderly males between the ages of 65 to 75 years
  2. Willingness to participate in the study
  3. Males without a chronic disease or acute illness that could affect protein and AA metabolism eg, diabetes, cancer, liver or kidney disease, HIV, acute cold or flu, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications.
  4. Males with hypertension if well controlled by medications

Exclusion Criteria:

1. Presence of disease known to affect protein and amino acids (AA) requirement and synthesis like diabetes, cancer, liver o kidney disease, HIV, acute cold or flu, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications.
2. On medications known to affect protein and amino acid metabolism like e.g. steroids.
3. Significant weight loss during the past month.
4. Individual on weight reducing diets.
5. Inability to tolerate the diet or unwilling to have blood drawn from a venous access for the purposes of the study.
6. Significant coffee consumption of more than 2 cups/day (400 mg of caffeine/day)
7. Significant Alcohol consumption of more than one drink/day ( 1 beer, ½ glass of wine)

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Urine (for measurement of 13C phenylalanine enrichment) and breath (for measurement of 13CO2 enrichment) samples will be collected on day 3 of the experiment between the 4th and 5th meal and after the 6th and 7th meal. | 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Rafii M, Chapman K, Elango R, Campbell WW, Ball RO, Pencharz PB, Courtney-Martin G. Dietary Protein Requirement of Men >65 Years Old Determined by the Indicator Amino Acid Oxidation Technique Is Higher than the Current Estimated Average Requirement. J Nutr. 2015 Apr 1;146(4):681-687. doi: 10.3945/jn.115.225631. PMID 26962173